CLINICAL TRIAL: NCT01049477
Title: The Effects of Music Therapy on Women's Anxiety Before and During Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMC 2007-0906
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2014-12

CONDITIONS: Pregnancy; Cesarean Section
Keywords: Pregnancy; Cesarean Section

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music therapy (Experimental): Experimental arm includes women undergoing cesarean section delivery listening to music before and after c/s. STAI will be completed pre and post operatively.
  Interventions: Other: Music group; Other: Non music group
- No music group (No Intervention): Subjects will not listen to music before and after c/s. STAI will be completed pre and post operatively.

INTERVENTIONS:
Other: Music group — The patients randomized to the music group of the study will listen to music 30 minutes in the holding room prior to their c/s. They will then listen to music after their c/s for 30 minutes. They will complete the STAI before and after their c/s.
  Arms: Music therapy
Other: Non music group — Patients randomized to the non music group will complete the STAI before and after their c/s, but not listen to music.
  Arms: Music therapy

SUMMARY:
The purpose of the study is to determine if listening to your choice of music with a portable mp3 player before and after a cesarean section for delivery of a baby will decrease the patient's anxiety level.

DETAILED DESCRIPTION:
Music has been suggested and evaluated as a therapeutic intervention to reduce preoperative anxiety for surgical patients. Music intervention in the immediate preoperative period may be effective in lowering anxiety levels during Cesarean delivery. If this investigation shows that music intervention before and after Cesarean delivery reduces anxiety levels, this intervention can be integrated into future operative care for women having scheduled or emergency Cesarean deliveries. Music therapy could be expanded to included patients undergoing other surgical procedures under regional anesthesia. The effect of reducing anxiety levels could aid in lactation initiation and improve infant bonding in new mothers, but it could also shorten postoperative recovery time for all surgical patients.

ELIGIBILITY:
Inclusion Criteria:Women age 18 and older with a history of one prior Cesarean delivery that are scheduled for a repeat Cesarean delivery under regional anesthesia, or women who are undergoing a primary cesarean section will be eligible to participate.

-

Exclusion Criteria:Women with cardiovascular disease, chronic hypertension, insulin dependent diabetes mellitus, multiple gestation pregnancies, psychiatric disorders, and fetal anomaly.

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The intervention of patient-selected music before and after Cesarean delivery will decrease anxiety levels in a patient population undergoing Cesarean delivery. | Before and after cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Heather Mertz, MD, Principal Investigator — Wake Forest University
Locations (1):
- Forsyth Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] 1. Gori F, Pasqualucci A, Corradetti F, et al. Maternal and neonatal outcome after cesarean section: The impact of anesthesia. The Journal of Maternal-Fetal and Neonatal Medicine 2007; 20(1):53-57. 2. Wang S, Kulkarni L, Dolev J, et al. Music and preoperative anxiety: A randomized, controlled study. Anesth Analg 2002; 94(6):1489-1494. 3. Chang S, Chen C. Effects of music therapy on women's physiologic measures, anxiety, and satisfaction during Cesarean delivery. Research in Nursing & Health 2005; 28:453-461. 4. Danhauer SC, Marler B, Rutherford CA, Lovato JF, et al. Music or guided imagery for women undergoing colposcopy: A randomized controlled study of effects on anxiety, perceived pain, and patient satisfaction. J low genit tract dis 2007; 11:39-45. 5. Yung PMB, Kam SC, Lau BWK, et al. The effect of music in managing preoperative stress for Chinese surgical patients in the operating room holding area: A controlled trial. International Journal of Stress Management 2003; 10(1):64-74. 6. Gaberson KB. The effect of humorous and musical distraction on preoperative anxiety. AORN Journal 1995; 62(5):784-791. 7. Pan P, Coghill R, Houle T, et al. Multifactorial and preoperative predictors for postcesarean section pain and analgesic requirement. Anesthesiology 2006; 104:417-425. 8. Maes M, Libbrecht I, Lin A, et al. Effects of pregnancy and delivery on serum prolyl endopeptidase (PEP) activity: alterations in serum PEP are related to increased anxiety in the early puerperium and to postpartum depression. Journal of Affective Disorders 2000; 57:125-137. 9. Zanardo V, Trevisanuto D, and Freato F. Maternal anxiety impairs lactation initiation and maintenance. Pediatrics 2006; 117:1859-1860. 10. Hundley V, Gurney E, Graham W, et al. Can anxiety in pregnant women be measured using the State-Trait Anxiety Inventory? Midwifery 1998; 14:118-121. 11. Man AKY, Yap JCM, Kwan SY, et al. The effect of intra-operative video on patient anxiety. Anesthesia 2003; 58:64-68.
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021